CLINICAL TRIAL: NCT03651557
Title: A Phase II, Double-blind, Randomized, Placebo-controlled, Multicenter Trial to Assess the Efficacy and Safety of Neu2000KWL in Patients Who Resuscitated After Out-of-hospital Cardiac Arrest Patient and Receiving Therapeutic Hypothermia
Brief Title: Antioxidant and NMDA Receptor Blocker Wins Anoxic Brain Damage of KorEa OHCA Patients
Acronym: AWAKE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: GNT Pharma (Industry)
Collaborators: Samsung Medical Center (Other); Chonnam National University Hospital (Other); Gangnam Severance Hospital (Other); Kyungpook National University Hospital (Other); Pusan National University Hospital (Other); Soonchunhyang University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Neu2000KWL-P02
Record Dates: First submitted 2018-07-26; First posted 2018-08-29 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2018-08

CONDITIONS: Cardiac Arrest
Keywords: Neu2000KWL; cerebral performance category; out-of-hospital cardiac arrest; neuroprotection; glutamate; N-Methyl-D-aspartate (NMDA) receptor antagonist; Anti-oxidant; free radical
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind (Subject, Caregiver, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neu2000KWL high dose (Experimental)
  Interventions: Drug: Neu2000KWL High-dose group
- Neu2000KWL low dose (Experimental)
  Interventions: Drug: Neu2000KWL Low-dose group
- saline (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neu2000KWL High-dose group — 1st infusion of 1500mg in patients within 4 hours following sudden cardiac arrest onset followed by 5 consecutive infusions of 750 mg at intervals of 12 hours(Total drug dosage is 5250mg.)
  Arms: Neu2000KWL high dose
Drug: Neu2000KWL Low-dose group — 1st infusion of 750mg in patients within 4 hours following sudden cardiac arrest onset followed by 5 consecutive infusions of 500 mg at intervals of 12 hours (Total drug dosage is 3250mg.)
  Arms: Neu2000KWL low dose
Drug: Placebo — 1st infusion of the same volume of saline in patients within 4 hours following sudden cardiac arrest onset followed by 5 consecutive infusions of the same volume of saline at intervals of 12 hours
  Arms: saline

SUMMARY:
This study aims to investigate the efficacy and safety of Neu2000KWL, a neuroprotectant, in patients resuscitated from out-of-hospital cardiac arrest and receiving therapeutic hypothermia.

DETAILED DESCRIPTION:
Lack of good neurological recovery is the biggest hurdle in the treatment of out-of-hospital cardia arrest. Neu2000KWL, a N-Methyl-D-aspartate (NMDA) receptor antagonist and an antioxidant, attenuated cerebral neuronal death and reduced hypoxic injury of brain in preclinical studies. Phase I clinical study has revealed that Neu2000KWL is very safe for treating human. In current study, the investigators will assess the efficacy of Neu2000KWL to compare the neurological biomarker, brain imaging, and clinical outcomes of patients successfully resuscitated from out-of-cardiac arrest treated by 3-day infusion of Neu2000KWL with patients assigned to placebo arm.

ELIGIBILITY:
Inclusion Criteria:

1. 19 Years to 80 Years (Adult)
2. Out-of-hospital cardiac arrest caused by non-perfusing cardiac rhythm
3. Successful resuscitation accompanied by ROSC time of more than 20 min
4. Therapeutic hypothermia is planned or initiated
5. The first infusion is planned within 4 hours after ROSC
6. Informed consent is obtained from patient or family member(s)
7. No concern with previous cardiovascular surgery

Exclusion Criteria:

1. Hypersensitivity to aspirin or sulfasalazine
2. Unwitnessed cardiac arrest
3. CPR time > 60 min
4. Therapeutic hypothermia is not planned
5. Use of extracorporeal membrane oxygenation (ECMO) at initiation of in-hospital resuscitation (E-CPR)
6. Very poor prognosis is expected: patients with (A) non-cardiac or respiratory arrest, (B) poor basal neurological status (C) secondary cardiac arrest caused by trauma, major bleeding, acute neurologic disease including stroke or tumor, (D) multiorgan failure or advanced malignancy
7. Pregnant or lactating women
8. Participated in other clinical studies within 90 days before randomization; or participating in other clinical trials at present
9. Intracranial bleeding verified by first brain CT imaging
10. The investigators consider the patients are not suitable for this trial

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Verification of difference between of Neuron specific enolase (NSE) value at after 4th infusion of Neu2000KWL. | The 3rd day of study (which corresponds to finished 4th infusion of Neu2000KWL).
  Blood concentration of neuron specific enolase (NSE)

SECONDARY OUTCOMES:
Verification of difference between the cumulative of neuron specific enolase (NSE) values at after 6th infusion of Neu2000KWL | The 4th day of study (which corresponds to finished 6th infusion of Neu2000KWL).
  Cumulative Blood concentration of neuron specific enolase (NSE)
Verification of the difference between groups of Change in NSE values at after the 2nd infusion of Neu2000KWL and after the 6th infusion | At the 24 hours and 72 hours after the first infusion of Neu2000KWL.
  The difference of blood neuron specific enolase (NSE) between 24 hour (day 1) and 72 hour (day 3) after the first infusion of Neu2000KWL.
Verification of difference between each group of NSE values at after 6th infusion after 1st infusion of Neu2000KWL and 24 hours after end of last infusion | The 4th and 5th day of study (which corresponds to the timepoint of finished treatment using Neu2000KWL and 24 hour after finished treatment using Neu2000KWL).
  The difference of blood neuron specific enolase (NSE) between day 4 and day 5
Verification of difference between the cerebral infarction at analysis of brain MRI's Apparent Diffusion Coefficient(ADC) images within 48 hours of the last infusion of Neu2000KWL | The 5th day of study (which corresponds to 48 hours after finished treatment using Neu2000KWL).
  Blood neuron specific enolase (NSE) at day 5
Verification of difference between groups of Neurological function evaluated by cerebral performance category (CPC) and modified Rankin Scale (mRS) at 5 day, 14 day, or discharge within 14 days, and 90 days after 1st infusion of Neu2000KWL. | 5 day, 14 day, or discharge within 14 days, and 90 days after 1st infusion of Neu2000KWL
  Neurological function evaluated by cerebral performance category (CPC), which ranges 1 to 5 (1: best, 5: worst), and neurological function evaluated by modified Rankin Scale (mRS), which ranges 0 to 6 (0:best, 6: worst)
Verification of difference between groups of Cumulative value of blood S100beta from 6th infusion after 1st infusion of Neu2000KWL. | The 4th day of study (which corresponds to finished 6th infusion of Neu2000KWL).
  Cumulative blood concentration of S100beta .

OTHER OUTCOMES:
Serious adverse event | 90 days
  Safety Outcome Measure
  Number of participants with treatment-related adverse events assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Mortality within 90 days | 90 days
  Safety Outcome Measure

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ho Choi, MD, Principal Investigator — Professor, Department of Emergency Medicine, Samsung Medical Center
Locations (6):
- South Korea (6):
  - Kyungpook National University Hospital, Daegu, Korea
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Pusan National University Hospital, Busan
  - Chonnam National University Hospital, Gwangju
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chun BJ, Yeom SR, Chung SP, Lee YH, Lee J, Kim YH, Lee JS, Lee JS, An CS, Gwag BJ, Choi JH. Nelonemdaz Treatment for Patients With Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. Crit Care Med. 2025 Apr 1;53(4):e772-e782. doi: 10.1097/CCM.0000000000006579. Epub 2025 Jan 14. PMID 39899673
- [Derived] Choi JH, Chun BJ, Yeom SR, Chung SP, Lee YH, Kim YH, Lee JS, Lee JH, Lee HG, Jin JY, An CS, Gwag BJ. Rationale and methods of the Antioxidant and NMDA receptor blocker Weans Anoxic brain damage of KorEa OHCA patients (AWAKE) trial. Trials. 2022 Jul 23;23(1):587. doi: 10.1186/s13063-022-06452-0. PMID 35871083